CLINICAL TRIAL: NCT06665412
Title: A Single-arm, Open-label, Multicenter, Investigator-led Observational Study to Evaluate the Efficacy and Safety of Dose Reduction of Radotinib as a First-line Treatment in Patients With Newly Diagnosed Chronic Phase Ph+ Chronic Myeloid Leukemia.
Brief Title: Efficacy and Safety of Dose Redution of Radotinib as a First Line Treament in Ph+ CML
Status: Recruiting | Type: Observational
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: RT51KR-IIT01
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Chronic Phase Ph+ Chronic Myeloid Leukemia
MeSH Terms: interventions — 4-methyl-N-(3-(4-methylimidazol-1-yl)-5-trifluoromethylphenyl)-3-(4-pyrazin-2-ylpyrimidin-2-ylamino)benzamide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Radotinib Hydrochloride — 200mg BID, every day up to 12months

SUMMARY:
The goal of this observational study is to learn about the efficacy and safety profile when Radotinib dose redution is performed in Ph+ CML subjects.

The main efficacy is checked by MMR rate by 12 months from IP treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 19 years old or older
2. Patients with confirmed diagnosis of chronic phase CML within last 8weeks(throung chromosome testing or bone marrow testing)

   * Chronic phase CML is defined as follows:

     * Blast in peripheral blood and bone marrow <15%

       * The sum of blast and promyelocyte in peripheral blood and bone marrow <30%

         * Basophil in peripheral blood <20%

           * Platelets count ≥ 50 × 109/L (≥ 50,000/mm3) (But, transient prior therapy related thrombocytopenia [<50 × 109/L (< 50,000/mm3)] is acceptable)

             * No extramedullary involvement other than enlargements of liver and spleen
3. Patients with positive Philadelphia chromosome and confirmed expression of BCR:ABL1 transcript
4. ECOG scale 0, 1 or 2
5. Patients who have adequate organ functions as defined below:

   * Total bilirubin < 1.5 × upper limit of normal (ULN)
   * SGOT and SGPT < 2.5× ULN
   * Creatinine < 1.5 × ULN
   * Serum amylase and lipase ≤ 1.5 × ULN
   * Alkaline Phosphatase ≤ 2.5 × ULN (only if not related to the tumor)
6. Women of childbearing potential should have a negative serum or urine pregnancy test
7. Women of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study and for a period of at least 1 month (4 weeks) after the last dose of investigational product in such a manner that the risk of pregnancy is minimized.
8. Patients providing written informed consent form before the study related screening procedures.

Exclusion Criteria:

1. Patients with Philadelphia chromosome negative
2. Patients who used Radotinib for 8 days or longer before study entry
3. Patients who had been treated with other targeted anti-cancer therapy, except for Hydrea or Agrylin, which inhibits the growth of leukemic cells
4. Patients who have hypersensitivity to active ingredient or any of the excipients of this investigational product.
5. Patients with impaired cardiac function as defined below:

   * Patients who cannot have QT intervals measured according to ECG

     * Complete left bundle branch block

       * Patients with cardiac pacemakers

         * Patients with congenital long QT syndrome or the family history of known long QT syndrome

           * The mean QTcF >450msec ECG tests at baseline

             * Clinically significant resting bradycardia (< 50 bpm) History of, or presence of symptomatic ventricular or atrial tachyarrhythmias

               * Clinically significant resting bradycardia (< 50 bpm)

                 * Medical history of clinically confirmed myocardial or infarctionof unstable angina (within last 12 months)

                   * Other clinically significant cardiac disease (e.g. congestive heart failure, or uncontrolled hypertension)
6. Cytologically confirmed CNS involvement (if asymptomatic, spinal fluid examination is not necessary prior to first treatment)
7. Severe or uncontrolled chronic medical condition (e.g., uncontrolled diabetes, active or uncontrolled infection)
8. Other significant congenital or acquired bleeding disorders that are not related to underlying leukemia
9. Patients who previously received radiotherapy to at least 25% of the bone marrow
10. Patients who had a major surgery within 4 weeks prior to study entry or has not recovered from side effects of such surgery
11. Patients who diagosed with another clinically significant malignant tumor wihin 5years before study etnry, excluding basal cell carcinoma
12. Patients who are currently receiving treatment with a strong CYP3A4 inhibitor (e.g., erythromycin, ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, ritonavir, mibefradil) or CYP3A4 inducer (e.g., dexamthasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbitol, St. John's Wort). Treatment cannot be safely discontinued or switched to a different medication prior to initiation of study treatment
13. Patients who are currently receiving treatment with a medication that has the potential to prolong the QT interval. Treatment cannot be safely discontinued or switched to a different medication prior to initiation of study treatment
14. Impairment of GI function or GI disease that may significantly alter absorption of study drugs (e.g., ulcerative colitis, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection, GI bypass surgery).
15. History of acute or chronic pancreatitis within last one year
16. Acute or chronic liver or pancreas disease or severe renal disease
17. Patients with HbsAg, HCV Ab positive

    * following subjects can be enrolled.

      * Inactive hepatitis B surface antigen (HBsAg) carriers(site specific local lab normal range lower limit assessed by investigator)
      * undergoding HCV Ab or HCV RNA testing judged by investigator to be eligible for enroll
18. History of HIV Ab positive or confirmed HIV Ab positvie.
19. Pregnant or the women with breast-feeding 2

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed, CP-CML patients
Sampling Method: Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate MMR rate up to 12months following the treatment of Radotinib | up to 12months

CONTACTS AND LOCATIONS:
Overall Officials: Na Yun Kim, Study Director — Il-Yang Pharm. Co., Ltd.
Locations (2):
- South Korea (2):
  - Hallym University Sacred Heart Hosptial, Anyang-si, Gyeonnggi-do
  - Keimyung University Daegu Dongsan Hospital, Daegu

IPD SHARING:
Plan to Share IPD: No